CLINICAL TRIAL: NCT06944119
Title: Assesment of the Immune Response to RSV Vaccine in Patients With Myeloma, Lymphoma and Hematological Leukemia
Status: Active, not recruiting | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0646-24-TLV
Record Dates: First submitted 2025-01-22; First posted 2025-04-25 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-04

CONDITIONS: Myeloma; Lymphoma; CLL; Myelodysplastic Syndrome; Leukemia Acute Myeloid - AML
MeSH Terms: conditions — Neoplasms, Plasma Cell; Lymphoma; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A prospective study in which hematological oncology patients who were vaccinated against RSV will undergo a blood test to assess their immune response to the vaccine. As part of the study, hematological oncology patients with CLL, lymphoma, acute leukemia, myelodysplastic syndrome, and multiple myeloma, who are being monitored at the Hematology Institute at Ichilov, will be offered a blood test to evaluate their immune response to the RSV vaccine (serology, neutralizing antibodies, and cellular response). In the study, a blood sample of up to 10 ml will be taken in a chemistry tube and blood bank on the day of vaccination and about one month after that. The serological test will be conducted in the hospital's virology laboratory. The test result and its significance will be communicated to the patient by the treating hematologist in TASMC clinic. In this group of patients, a follow-up will be conducted over a 12-month period (during routine clinic visits) to document the incidence of RSV infection and complications related to the vaccine.

DETAILED DESCRIPTION:
participants 250 Single-center Research hypothesis approximately 60%-70% of the 250 hematological oncology patients who will participate in the study will achieve a positive serological response. This estimate is based on a study published in the NEJM which included participants aged 60 and above, without hematological oncological diseases or other conditions causing immunosuppression, where a response was observed in 83.7% of participants. the investigators estimate that the response rate in hematological oncology patients will be lower, ranging from 60-70%, reflecting the degree of immune suppression associated with their disease and the treatment they received.

The study will include patients with chronic lymphocytic leukemia (CLL), lymphoma, myelodysplastic syndrome, leukemia, and myeloma. The investigatorsexpect that approximately 60 patients will belong to each of these subgroups, so the sample size will allow an assessment of the immune response within these subpopulations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 years and older
* Patients diagnosed with multiple myeloma(MM) or lymphoma or CLL or myelodysplastic syndrome (MDS) or acute leukemia

Exclusion Criteria:

* Patients who have been previously vaccinated against RSV
* Patients who have experienced a severe reaction to any vaccine in the past

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 60 years and older diagnosed with multiple myeloma, lymphoma, CLL, myelodysplastic syndrome, and acute leukemia who are scheduled to receive the RSV vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
To assess the immune response to the RSV vaccine in patients with CLL, multiple myeloma, lymphoma, myelodysplastic syndrome, and acute leukemia, by measuring antibody levels in the blood up to 6 weeks after receiving the vaccine | Up to 45 days post-vaccination
  The response rate Is expected to be 60-70%

SECONDARY OUTCOMES:
To evaluate the safety of the vaccine by measuring the incidence of Treatment-Emergent Adverse Events | Up to 45 days post-vaccination
  The safety of the vaccine will be evaluated in hemato-oncological patients through the collection of adverse events (AEs) and serious adverse events (SAEs) up to 45 days post-vaccination.
To identify factors predicting success/failure in achieving an antibody response to the vaccine. | Up to 1 year
  1. All adverse events occurring within 30 days following vaccination.
  2. Grade≥3 adverse events occurring within 30 days following vaccination.
To assess the incidence rate of RSV infection in individuals vaccinated against RSV over a 12-month period following vaccination. | Up to 1 year
  We will assess the incidence rate of RSV infection in individuals vaccinated against RSV over a 12-month period by collecting data on RSV infections during the year following vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Irit Avivi, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No